CLINICAL TRIAL: NCT05500651
Title: The Effect of Dance and Movement Therapy as a Group Work Technique on Negative Symptoms and Disability in Patients With Schizophrenia
Brief Title: Dance and Movement Therapy in Patients With Schizophrenia
Acronym: DMTinSchizo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Gonca Ustun, Assist. Prof., Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AmasyaU8
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia; Negative Symptoms in Schizophrenia; Disabilities Mental; Dance Therapy
Keywords: Dance and movement therapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: A repetitive measure design with a pretest-posttest control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Dance and movement therapy is planned to be applied once a week as a total of 12 sessions of 60 minutes. First session; meeting, warming up, determining the group rules, explaining the principles, determining the expectations activities. Subsequent sessions; The greeting is completed with warm-up, initiation, continuation and closing activities. During the warm-up phase, the whole group comes together to form a circle, generally standing, in order to ensure the group dynamic. It starts with simple warm-up exercises such as breathing and muscle relaxation and continues with body awareness exercises. In the continuation (development of themes) stage, practices are included according to the characteristics and needs of the group.
  Interventions: Other: Dance and Movement Therapy (DMT)
- Control group (No Intervention)

INTERVENTIONS:
Other: Dance and Movement Therapy (DMT) — Dance and movement therapy is planned to be applied once a week as a total of 12 sessions of 60 minutes. First session; meeting, warming up, determining the group rules, explaining the principles, determining the expectations activities. Subsequent sessions; The greeting is completed with warm-up, initiation, continuation and closing activities. During the warm-up phase, the whole group comes together to form a circle, generally standing, in order to ensure the group dynamic. It starts with simple warm-up exercises such as breathing and muscle relaxation and continues with body awareness exercises. In the continuation (development of themes) stage, practices are included according to the characteristics and needs of the group.
  Arms: Experimental group

SUMMARY:
Introduction: Schizophrenia is a mental disorder that starts at a young age and progresses with positive (hallucination, delusion) and negative (decreased emotional participation, reluctance) symptoms. While drug therapy in schizophrenia targets positive symptoms; psychotherapies are needed in the treatment of negative symptoms. It is seen that especially art therapies such as occupational and music support recovery and rehabilitation. In addition, it is stated that dance and movement therapy is effective in ensuring social participation of patients. There are a limited number of studies demonstrating the effect of dance and movement therapy on schizophrenia patients.

Aim: This project was planned to examine the effects of dance and movement therapy techniques to be applied to patients with schizophrenia on patients' negative symptoms and disability.

Method: In this project, which was planned in a repetitive measure design with a pretest-posttest control group, dance and movement therapy techniques, consisting of 12 sessions in total, will be applied to schizophrenic patients in a Community Mental Health Center once a week. Negative symptoms and disability levels will be determined before, after and a month after the application. The findings obtained as a result of these three follow-ups will be evaluated.

Project Outputs: Reduction of negative symptoms and disability will enable schizophrenic patients to become individuals who can express themselves better in their family and society and have an increased quality of life. It is thought that these gains will increase patients' compliance with treatment, prevent recurrent symptoms and reduce hospitalizations. The results will also constitute a scientific source for the studies to be carried out in the field.

ELIGIBILITY:
Inclusion Criteria:

* have been diagnosed with schizophrenia for at least two years
* not have been hospitalized in the past 3 months

Exclusion Criteria:

* have a therapy/psychoeducation program that they attend regularly
* have a known physical or neurological disease
* having just started the Community Mental Health Center

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
The Scale for the Assessment of Negative Symptoms (SANS) | 6 months
  Scale; It consists of five parts, including flattening or blunting in affect, alogy, decreased energy and desire, lack of pleasure and social withdrawal, attention, and a total of 24 items. Scale items 0=none; 1=doubtful; 2=light; 3=medium; 4=pronounced; It is scored as 5=severe. The negative symptoms rating scale is a type of scale that the interviewer evaluates. The filling of the scale is based on the interview with the patient, the observations during the interview and the information received from the people around the patient. Cronbach's alpha for the whole scale is 0.94.
  Values that can be taken from the Scale for the Assessment of Negative Symptoms (SANS); minimum=0, maximum=120 points. It shows that as the score increases, the severity of negative symptoms increases.
Disability Evaluation Schedule (WHO-DAS-II) | 6 months
  Disability Assessment Chart is a 36-item scale. This tool tries to determine how much difficulty an individual with schizophrenia has while performing certain activities and consists of 6 areas that include activities that are considered important in many cultures. These are grouped under the headings of understanding and communicating, moving and moving from place to place, self-care, human relations, life activities, participation in social life. In questions about all these areas, it is asked how much difficulty the person has had during that activity in the last month, and the answers received as not at all, mild, moderate, very much, excessively/not at all are scored between 1-5. It is applied by the interviewer in approximately 20 minutes. Cronbach's alpha for the whole scale is 0.92.
  Values that can be taken from the Disability Evaluation Schedule (WHO-DAS-II); minimum=0, maximum=100 points. It shows that as the score increases, the severity of disability increases.

OTHER OUTCOMES:
Personal Information Form | 2 weeks
  The questionnaire form prepared by the project team consists of 10 questions in total, including the socio-demographic characteristics (age, gender, marital status, education level, employment status, income level, cohabitants) of the patients and their disease-related characteristics (age of onset of disease, duration of disease (years), number of hospitalizations).

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya Üniversitesi Sabuncuoğlu Şerefeddin Eğitim Ve Araştirma Hastanesi, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No